CLINICAL TRIAL: NCT07343466
Title: Klinische Studie Zur Untersuchung Der Lebensqualität Und Des Einflusses Von Stress Auf Den Postoperativen Verlauf Von Patienten Nach Device-Implantation
Brief Title: Quality of Life and the Influence of Stress on the Postoperative Course of Patients After Device Implantation
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 24-12310-BO
Record Dates: First submitted 2025-08-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Quality of Life (QOL) and Impact of Stress
Keywords: Impact of Stress; postoperative course; ICD; CRT; Pacemaker; Event-Recorder; prospektive; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with indication for device implantation (pacemaker, ICD, CRT, event recorder): Patients with cardiac diseases, that makes a device implantation (pacemaker, ICD, CRT, event recorder) necessary, including primary and secondary indication for an ICD.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — survery over 36 months with comparison of the questionnares with risk-factors, blood-samples and physical fitness of the patient

SUMMARY:
The project "Investigating Quality of Life and the Influence of Stress on the Postoperative Course of Patients After Device Implantation" aims to investigate the relationship between stress and the postoperative healing process of patients who have had a medical device implanted. These devices include pacemakers for the treatment of bradycardia, implantable cardioverter-defibrillators (ICDs) for the treatment of tachycardia in primary and secondary prevention, and cardiac resynchronization therapy (CRT) devices and event recorders. The study will analyze the influence of stress on the postoperative course, potential complications, and overall quality of life. A combination of medical examinations and surveys will be used to analyze how psychological stress influences the physical healing process and which measures can contribute to improving quality of life and treatment success. The surgical procedure for implanting devices is not part of the study; this is an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal capacity with an indication for device implantation (pacemaker, ICD, CRT, event recorder) who present at the Department of Cardiology and Angiology at the University Hospital Essen and consent to participate in the study will be included.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for device implantation (pacemaker, ICD, CRT, event recorder) who present at the Department of Cardiology and Angiology at the University Hospital Essen
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of device-related complications | 36 Months
  Measures the incidence of device-related complications, this includes: Complications related to Device- pockets, leads and infections connected to the devices

SECONDARY OUTCOMES:
hospitalisation rate | 36 Months
  Analyzes how often and when the Patient got hospitalized
Number of participants with the following arrhythmic events: ventrikular tachykardia and ventrikular fibrillation | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  Following device implantation, subsequent follow-up evaluations include device interrogation to assess stored arrhythmic events. Specifically, the analysis focuses on the detection of ventricular tachycardia and ventricular fibrillation. The frequency of these arrhythmias is systematically recorded for each study participant.
Changes in functional capacity | Baseline (at 4-6 weeks) , after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  changes in functional capacity will be recorded using the established 6-minute walk test. The unit of measurement for the distance covered in 6 minutes will be meters.
combined global stress measure | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The outcome is based on a published RCT in Circulation by Blumenthal et al. . A global stress measure (mean rank), was the primary outcome combining the following components at baseline and following treatment: Beck Depression Inventory II, Spielberger Anxiety Inventory-State, General Health Questionnaire, PROMIS Anger Questionnaire, and Perceived Stress Scale. A range from 1 to 147 was present with higher scores suggestive of better function. The change in each individual scaled score is presented in secondary outcome. (see also NCT00981253)
Health-related quality of life - SF-36 | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The investigators will apply the Short Form-36 health questionnaire [36,37]. The SF-36 is an eight-dimensional scale consisting of 36 items. It assesses health-related quality of life based on physical, social, and psychological functioning, role behavior due to physical and psychological functional impairment, physical pain, general health perception, and vitality.
Health-related Quality of life - EQ-5D-5L | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The investigators will apply the European Quality of Life 5 Dimensions 5 Level survey (EQ-5D-5L) [36,37]. The EQ-5D-5L consists of five health-related dimensions that can be assessed at five levels.
Health-related Quality of life - VAS for general health | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The questionnaire contains a visual analog scale for assessing general health. It consists of a straight line from 0 to 100, with endpoints representing extreme values-such as "worst imaginable health" on one side and "best imaginable health" on the other. The participants mark a position on the line. The position of the mark provides a numerical value.
Depression symptoms (BDI-II) | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The BDI-II is a self-report questionnaire comprising 21 items that assess depression severity. Its reliability and validity have been established through various studies among diverse populations and cultural backgrounds. Higher scores indicates increased depression symptoms
Anxiety symptoms (STAI) | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The STAI is the most authoritative tool for assessing anxiety in adults, precisely distinguishing between transient "state anxiety" and persistent "trait anxiety". The STAI measures anxiety with 20 items and has a range of 20 to 80. A higher score indicates more pronounced anxiety
PROMIS-Anger Scale | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The PROMIS Anger scale comprises eight items that evaluate various aspects of anger. Scores on the scale range from 8 to 40, with higher scores indicating greater levels of anger
GHQ, Evaluation of distress | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The GHQ assesses general distress and consists of 12 items. Respondents' scores range from 0 to 36, where higher scores correspond to increased distress
Perceived Stress Scale | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  The Perceived Stress Scale-10 item version is a short tool for the assessment of how individuals perceive stress in their lives. The values range from 0 to 40. Higher values indicate higher perceived stress.
Appropriate vs. inappropriate Shocks | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  All ICD shock events occurring during the follow-up period will be classified as either appropriate or inappropriate, based on predefined criteria.
  Appropriate shocks will be defined as those delivered in response to documented, life-threatening ventricular arrhythmias, including:
  * Ventricular tachycardia (VT)
  * Ventricular fibrillation (VF),
  Inappropriate shocks will be defined as those delivered in the absence of a qualifying ventricular arrhythmia. For example:
  -Supraventricular tachycardias (e.g., atrial fibrillation or flutter) misclassified as VT/VF or Oversensing due to lead malfunction, signal noise, or double counting.
  All shock events will be reviewed using intracardiac electrograms and device event logs retrieved from the ICD or CRT-D memory. When available, surface ECG data will be used to support rhythm interpretation.
  A shock will only be classified as appropriate if there is clear evidence of a ventricular arrythmia
proinflammatory mediators- IL6 | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  IL-6 is measured in pg/ml. Standard value is under 4.4 pg/ml. Higher values indicate an increased stress level
Proinflammatory mediators - CRP | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  C-reactive protein (CRP) is measured in mg/dl. Standard value is under 0.5 mg/dl. Higher values indicate an increased stress level.
Proinflammatory mediators- PCT | Baseline, after 4-6 weeks, after 6 months, after 12 months, after 18 months, after 24 months, after 30 months, after 36 months
  Procalcitonin is measured in ng/ml. Standard value is under 0.5 ng/ml. Higher values correlate with systemic inflammatory reaction and indicate bacterial infections.

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, Univ.-Prof. Dr. med., Study Chair — Universitätsklinikum Essen; Julia Lortz, Prof. Dr. med., Study Director — Universitätsklinikum Essen; Muhammed Kurt, Dr. med., Study Director — Universitätsklinikum Essen
Locations (1):
- Universitätsklinikum Essen, Klinik für Kardiologie und Angiologie, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
All collected data will be stored in pseudonymized form and retained for 10 years after completion or termination of the study, after which it will be destroyed. All study documents, including the pseudonymized list, will be stored and managed on the clinic's own servers. Access to data storage and management will be restricted to authorized personnel (study management, relevant study physicians, and medical doctoral students). Data will not be shared with third parties.

REFERENCES:
- [Background] Golbidi S, Frisbee JC, Laher I. Chronic stress impacts the cardiovascular system: animal models and clinical outcomes. Am J Physiol Heart Circ Physiol. 2015 Jun 15;308(12):H1476-98. doi: 10.1152/ajpheart.00859.2014. Epub 2015 Apr 17. PMID 25888514
- [Background] Pedersen SS, Wehberg S, Nielsen JC, Riahi S, Larroude C, Philbert BT, Johansen JB; DEFIB-WOMEN Investigators. Patients with an implantable cardioverter defibrillator at risk of poorer psychological health during 24 months of follow-up (results from the Danish national DEFIB-WOMEN study). Gen Hosp Psychiatry. 2023 Jan-Feb;80:54-61. doi: 10.1016/j.genhosppsych.2022.12.006. Epub 2023 Jan 3. PMID 36638700
- [Background] Kim J, Park JK, Choi J, Kim SH, On YK, Shin MS, Choi N, Heo S. Changes in the Physical Function and Psychological Distress from Pre-Implant to 1, 6, and 12 Months Post-Implant in Patients Undergoing Implantable Cardioverter Defibrillator Therapy. J Clin Med. 2020 Jan 22;9(2):307. doi: 10.3390/jcm9020307. PMID 31979074
- [Background] van Barreveld M, Verstraelen TE, van Dessel PFHM, Boersma LVA, Delnoy PPHM, Tuinenburg AE, Theuns DAMJ, van der Voort PH, Kimman GJ, Buskens E, Zwinderman AH, Wilde AAM, Dijkgraaf MGW; DO-IT Registry Investigators. Dutch Outcome in Implantable Cardioverter-Defibrillator Therapy: Implantable Cardioverter-Defibrillator-Related Complications in a Contemporary Primary Prevention Cohort. J Am Heart Assoc. 2021 Apr 6;10(7):e018063. doi: 10.1161/JAHA.120.018063. Epub 2021 Mar 31. PMID 33787324
- [Background] Miller JL, Thylen I, Elayi SC, Etaee F, Fleming S, Czarapata MM, Lennie TA, Moser DK. Multi-morbidity burden, psychological distress, and quality of life in implantable cardioverter defibrillator recipients: Results from a nationwide study. J Psychosom Res. 2019 May;120:39-45. doi: 10.1016/j.jpsychores.2019.03.006. Epub 2019 Mar 5. PMID 30929706
- [Background] Lampert R. Managing with pacemakers and implantable cardioverter defibrillators. Circulation. 2013 Oct 1;128(14):1576-85. doi: 10.1161/CIRCULATIONAHA.113.001555. No abstract available. PMID 24081953
- [Background] Linde C. Quality-of-life in pacemaker and implantable cardioverter defibrillator recipients. Pacing Clin Electrophysiol. 2000 Jun;23(6):931-3. doi: 10.1111/j.1540-8159.2000.tb00876.x. No abstract available. PMID 10879374
- [Background] Su SF, Wu MS. Arrhythmia Perception and Quality of Life in Bradyarrhythmia Patients Following Permanent Pacemaker Implantation. Clin Nurs Res. 2021 Feb;30(2):183-192. doi: 10.1177/1054773819880297. Epub 2019 Oct 16. PMID 31617405
- [Background] Sikora K, Wawryniuk A, Luczyk RJ, Sawicka K, Zwolak A. The Occurrence of Stress, Illness Acceptance and the Quality of Life of Patients after Pacemaker Implantation. Int J Environ Res Public Health. 2022 Oct 29;19(21):14133. doi: 10.3390/ijerph192114133. PMID 36361008
- [Background] Iliou MC, Blanchard JC, Lamar-Tanguy A, Cristofini P, Ledru F. Cardiac rehabilitation in patients with pacemakers and implantable cardioverter defibrillators. Monaldi Arch Chest Dis. 2016 Oct 14;86(1-2):756. doi: 10.4081/monaldi.2016.756. PMID 27748467